CLINICAL TRIAL: NCT01261208
Title: The Study of the Prevalence of Helicobacter Pylori Infection Among HIV/AIDS Cohort
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-990152
Record Dates: First submitted 2010-07-08; First posted 2010-12-16 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2017-01

CONDITIONS: HIV
Keywords: HIV, AIDS, Helicobacter pylori
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Study is to investigate the prevalence of Helicobacter Pylori infection among the HIV/AIDS group. The study will screen the patients who were confirmed HIV/AIDS in Kaohsiung Medical University Hospital and collect the cases who were suspicious of Helicobacter Pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of HIV
* the person who have stomach pain, vomiting or nausea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV/AIDS group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
all cause stomach pain | six months

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Tropical medicine center, Kaohsiung City, Taiwan